CLINICAL TRIAL: NCT06182007
Title: Pneumothorax After Cardiopulmonary Resuscitation Following Out-of-Hospital Cardiac Arrest - Analysis of Incidence, Risk Factors and Impact on Outcome
Brief Title: Post-Resuscitation Pneumothorax - Analysis of Incidence, Risk Factors and Outcome Relevance
Status: Completed | Type: Observational
Sponsor: Auinger, Daniel MD (Other)
Responsible Party: Sponsor-Investigator, Auinger, Daniel MD, MD, Medical University of Graz
Organization: Medical University of Graz (Other)
Other Study IDs: PostCPRptx
Record Dates: First submitted 2023-12-04; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Cardiac Arrest; Pneumothorax; Resuscitation
MeSH Terms: conditions — Heart Arrest; Pneumothorax | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No Pneumothorax: Patients with no pneumothorax reported from the first chest imaging after hospital admission.
  Interventions: Procedure: Cardiopulmonary Resuscitation
- Pneumothorax: Patients with a pneumothorax reported from the first chest imaging after hospital admission.
  Interventions: Procedure: Cardiopulmonary Resuscitation

INTERVENTIONS:
Procedure: Cardiopulmonary Resuscitation — Cardiopulmonary Resuscitation (Advanced Life Support) according to current guidelines

SUMMARY:
In this retrospective study, the investigators seek to investigate the incidence of pneumothorax following possible risk factors, and elucidate its association with outcomes.

DETAILED DESCRIPTION:
This is a retrospective analysis of routine data, collected by a single Emergency Medical System (EMS). Adult patients (≥18 years) hospitalised after Out-of-Hospital Cardiac Arrest (OHCA) who received chest compressions and underwent chest imaging within 12 hours after hospital admission were included.

Variables and outcomes ascertained are built up of the core elements of the latest version of the Utstein Resuscitation Registry Template for OHCA. This includes sex, age, aetiology of arrest, response times of the first emergency medical service team and emergency physician, witnessed cardiac arrest, bystander CPR/AED, arrest location, first monitored rhythm, defibrillation time, drugs given, reperfusion attempted and target temperature management. Additional variables studied were pre-existing health status represented by the Pre Emergency Status Assessment (PESA), history of lung disease, no-flow-time (time from collapse until initiation of CPR), use of a mechanical chest compression device and prehospital CPR duration.

The primary outcome is incidence of pneumothorax, secondary outcomes are survival to hospital discharge and favourable neurological condition at hospital discharge defined by a cerebral performance category (CPC) of 1 or 2.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized after out of hospital cardiac arrest
* Chest compressions received
* Chest imaging within the first 12 hours of admission

Exclusion Criteria:

* Traumatic cardiac arrest
* Chest trauma/surgery/pneumothorax one month prior to cardiac arrest

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Mid-Size European city + surrounding areas
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Presence of pneumothorax | within 12 hours of admission

SECONDARY OUTCOMES:
Survival | to hospital discharge (up to 2 months)
Cerebral Performance Category | at hospital discharge (up to 2 months)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Prause, Prof., Study Director — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Auinger D, Hotzer D, Zajic P, Orlob S, Heschl S, Fida S, Zoidl P, Honnef G, Friedl H, Smolle-Juttner FM, Prause G. Post-resuscitation pneumothorax: retrospective analysis of incidence, risk factors and outcome-relevance. Scand J Trauma Resusc Emerg Med. 2024 Sep 5;32(1):82. doi: 10.1186/s13049-024-01260-8. PMID 39238051